CLINICAL TRIAL: NCT06473883
Title: Effects of Vestibulo-oculomotor and Neuromuscular Training on the Incidence of Concussions and Musculoskeletal Injuries in Competitive Female Football Players
Brief Title: The Impact of Eye and Body Training on the Injury Rate of Concussions in Female Soccer Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BrainCare Medical Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20240126
Record Dates: First submitted 2024-06-03; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Concussion, Brain; Musculoskeletal Pain
MeSH Terms: conditions — Brain Concussion; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training recommendation (Experimental): The intervention group will receive training recommendations to prevent concussions and other injuries and improve their performance.
  Interventions: Other: Training recommendation
- Normal training (No Intervention): The control group will continue with their regular training without any recommendations for the prevention of head injuries.

INTERVENTIONS:
Other: Training recommendation — The players in the intervention group are also given specific training recommendations for the prevention of head injuries, which are compiled by experts (sports scientists, physiotherapists and neuroscientists). The exercise selection covers several areas that can be affected after a head injury. Each section contains 8 different exercises with increasing levels of difficulty (3x Basic-3x Intermediate-2x Advanced). The recommendations should be used as a warm-up program throughout the season before each training session. The coach or athletic coach will lead the warm-up program and ensure that each player follows the sequence and completes each phase according to the scheduled weeks. The warm-up program should be conducted as an 8-week cycle.
  Arms: Training recommendation

SUMMARY:
The research project aims to find out how special training influences the frequency and severity of injuries among female footballers in the top Swiss league. The project also aims to help establish normative values that are specifically tailored to women. The participating clubs will be randomly assigned to a comprehensive pre-season baseline examination with training recommendations based on the performed examinations (intervention group) or control group (normal training). Over the course of the 2024/2025 season, both groups will be compared in terms of the incidence and severity of concussions and musculoskeletal injuries. Initial results will be available in spring 2025 to coincide with the start of the European Women's Football Championship.

The investigators' hypothesis is that the training recommendations in the intervention group will lead to a lower incidence of concussions and that the players will show better injury prevention as a result of these exercises.

DETAILED DESCRIPTION:
All clubs in the top women's league in football will be contacted and asked to take part in the study. The baseline examinations will ideally take place in June and August 2024 to allow sufficient time to implement the training recommendations. The baseline examinations include a range of assessments addressing various systems potentially impacted by a concussion. These assessments encompass a standardized questionnaire, as well as vestibular, neurocognitive, balance, neck, and neurological evaluations.

Due to the availability of the players, baseline examinations may also have to take place in September. The players in the intervention group are also given specific training recommendations for the prevention of head injuries, which are compiled by experts (neurologists, sports scientists, physiotherapists and neuroscientists). The exercise selection covers several areas that can be affected after a head injury. Each section contains 8 different exercises with increasing levels of difficulty (3x Basic-3x Intermediate-2x Advanced). The recommendations should be used as a warm-up program throughout the season before each training session. The coach or athletic coach will lead the warm-up program and ensure that each player follows the sequence and completes each phase according to the scheduled weeks. The warm-up program should be conducted as an 8-week cycle.

The exercises are sent to the coaching staff in writing and by means of a video using our Neuroreha-Tool app. The coaches have access to the specific prescribed exercises. Each exercise is repeated 2-3 times and each exercise takes 50 seconds. In total, the warm-up will take 10-15 minutes.

During the football season from August 2024 to April 2025, players (both intervention and control groups) will be asked every two weeks to submit information about any injuries sustained in the match via the My REDCap app or the REDCap online survey. In the event of an injury, the date, type, and injured body region will be recorded via REDCap. Training adherence will also be documented for both groups (intervention group: number of training minutes for specific vestibulo-oculomotor and/or neuromuscular training exercises; control group: minutes of regular training).

After 8 weeks, a follow-up of the standard baseline tests will be repeated to measure the effects of the training recommendations. Each player receives a short report on the results of their examination within one week of the follow-up examination.

If a player suffers a concussion, they will be asked to complete the post-concussion symptom scale (PCSS). Players can also indicate if they wish to be contacted by the BrainCare institute for targeted diagnostics and/or therapy. On the day of the baseline examination, players will be thoroughly informed about the definition and correct recording of all endpoints collected in the follow-up. This information will also be available online on the app at any time. A recently published study confirms the usefulness and user-friendliness of a mobile app for monitoring training adherence and assessing pain using a pain rating scale.

Once a month, the club's contact person - ideally a member of the medical team who was also present at the baseline test - is contacted by the project management to verify the information and record the severity (i.e. the number of days the player is out of action) of injuries. The number of match appearances played (in hours) is determined using Power BI from the Swiss Football Association (football.ch).

ELIGIBILITY:
Inclusion Criteria:

* Registered player for a club in the top Swiss soccer league
* No symptoms of acute head injury at the start of the study
* Sufficient language skills to understand the study information and the informed consent form and to answer questionnaires and anamnestic questions correctly.

Exclusion Criteria:

* Symptomatic chronic diseases (e.g. tumor diseases, diabetes mellitus, cardiovascular diseases) with the exception of osteoarthritis and controlled (normotensively controlled) arterial hypertension
* Pregnancy
* Diagnosis of a psychiatric disorder/disease
* Drug abuse
* For the neuropsychological test: Known learning disability/disorder

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of injury frequency | 1 year
  Injury frequency will be gauged via REDCap questionnaires, capturing date, type, and injured region. Training adherence will be noted: the intervention group reports specific vestibulo-oculomotor and/or neuromuscular exercise minutes, while the control group reports normal training minutes. Concussed players complete the Post-Concussion Symptom Scale (PCSS). The PCSS is designed to quantify the range and severity of symptoms that can occur after a concussion. It helps healthcare professionals monitor changes in symptoms over time and make informed decisions about an individual's recovery and readiness to return to activities.Each symptom is rated on a scale, typically from 0 to 6, where 0 means the symptom is not present and 5-6 indicates severe severity.
  Questionnaires occur at baseline, 8-week follow-up, and biweekly until season end for all players.

SECONDARY OUTCOMES:
Clinical cervical spine/jaw exam: | 1 year
  The examination of the cervical spine and the surrounding tissue is used to identify cervical causes of headaches. Assessments include range of motion (degrees) and isometric strength (N) for the cervical spine, and extent of movement and deviation of mouth opening (degrees) for the jaw.
Video-Head Impulse Test (vHIT) | 1 year
  Passive, fast and low-amplitude rotational movements (head impulses, 10-15° eccentricity) are performed in the planes of each pair of semicircular canals (horizontal, RALP (right front-left rear), LARP (left front-right rear)) and induce VOR responses. During the examination, the subject is asked to fixate a target straight ahead. The eye movements during the VOR are measured with a high-speed video camera.
  Evaluation of gain (ratio between head and eye movement) and presence of saccades (rapid, corrective eye movements) are measured.
Dynamic Visual Acuity (DVA) | 1 year
  During the DVA, visual acuity is determined during head movements in order to measure the effectiveness of the visual stabilization function. Static visual acuity (visual acuity without head movement) is determined by reducing the size of a Landolt with C on a computer screen until the athlete is no longer able to read it correctly. The visual acuity is then obtained with head movements (120°/s, ±30°). If the difference between the static and dynamic visual acuity is more than 0.2 logMAR, there is a visual stabilization disorder.The difference between static and dynamic visual acuity is assessed in logMAR.
Vestibulo/Oculomotor Screening (VOMS) | 1 year
  The VOMS tests eye movements and vestibulo-oculomotor coordination. The screening covers five areas: Smooth pursuit, horizontal and vertical saccades, near convergence distance, horizontal vestibular eye reflex and visual motion sensitivity. For each area, the symptoms are rated on a Visual analogue scale (VAS), typically from 0 to 10, where 0 means the symptom is not present and 8-10 indicates severe severity. The near point convergence distance is measured in centimeters (cm).
Modified Balance Error Scoring System-Test (BESS) | 1 year
  BESS is a reliable and inexpensive tool to measure static balance. BESS consists of 6 tests that include both leg stance, one leg stance and tandem stance conditions, respectively, on both hard and foam surfaces with eyes closed. A stopwatch is used to determine participants' time during 20-second stance tests. The grading method is based on the score of the error table in the six tests. Errors include lifting the hip, walking, opening the eyes, grasping something, falling, leaving the test position after 5 seconds, flexion or abduction of the upper leg more than 30 degrees, and lifting the heel or front of the leg on the surface. If more than one mistake is made at the same time, they are counted as one mistake. The maximum total number of errors for any test is taken to be 10 (a higher score indicates mor balance errors and greater balance impairment).
Dual Task - Concussion Balance Test (COBALT) | 1 year
  The COBALT assesses balance through 5 conditions: 1 single-task and 4 dual-task. Participants are timed for 20 seconds using a stopwatch. In the single-task, they count backwards by 7s from 100. Dual-task conditions combine balance exercises with the cognitive task, with and without foam:
  1. Double leg stance with eyes closed, head rotating side to side to a metronome at 120 bpm.
  2. Eyes open, arms outstretched, thumbs up, focusing on thumbs while rotating side to side to a metronome at 40 bpm.
  Scoring uses an error table across conditions. Errors include cognitive mistakes, hip lifting, walking, eye opening, grasping, falling, leaving position early, leg movement beyond 30 degrees, and not syncing head or trunk rotation with the metronome. Each test's maximum errors are 10, with higher scores indicating more balance issues and impairment.
Postural Control - Sway path length | 1 year
  Sway path length measurement using an accelerometer involves tracking the movement of the center of pressure (COP) during the BESS and COBALT. This measure provides an objective assessment of postural control by quantifying the total distance the COP travels. An accelerometer is placed on the hip to capture the body's movements, and the data is analyzed using specialized balance software. The sway path length is measured in millimeters (mm).
Postural Control - sway path velocity | 1 year
  Sway path velocity measurement involves quantifying the speed at which the center of pressure (COP) moves. This parameter provides an objective assessment of postural control by indicating how quickly the COP travels. An accelerometer is placed on the hip to capture the body's movements, and the data is analyzed using specialized balance software. The measure is performed during the BESS and COBALT. The sway path velocity is measured in millimeters per seconds (mm/s).
Latency in horizontal saccades | 1 year
  Saccade latency in milliseconds (ms) during horizontal paradigms. The participant sits in front of a computer screen displaying a moving symbol, which they must follow without moving their head. Eye movements are recorded and analyzed using an eye-tracking device.
Latency in vertical saccades | 1 year
  Saccade latency in milliseconds (ms) during vertical paradigms. The participant sits in front of a computer screen displaying a moving symbol, which they must follow without moving their head. Eye movements are recorded and analyzed using an eye-tracking device.
Velocity in horizontal saccades | 1 year
  Saccade velocity in degrees per seconds (˚/s) during horizontal paradigms. The participant sits in front of a computer screen displaying a moving symbol, which they must follow without moving their head. Eye movements are recorded and analyzed using an eye-tracking device.
Velocity in vertical saccades | 1 year
  Saccade velocity in degrees per seconds (˚/s) during vertical paradigms. The participant sits in front of a computer screen displaying a moving symbol, which they must follow without moving their head. Eye movements are recorded and analyzed using an eye-tracking device.
Horizontal smooth pursuit gain | 1 year
  The gain refers to the accuracy with which the eyes match the velocity of a moving target. It is a measure of how well the eye movement system keeps up with the speed of the moving object in the horizontal plane. Specifically, gain is calculated as the ratio of eye movement velocity to target velocity. The participant sits in front of a computer screen displaying a moving symbol, which they must follow without moving their head. Eye movements are recorded and analyzed using an eye-tracking device.
Vertical smooth pursuit gain | 1 year
  The gain refers to the accuracy with which the eyes match the velocity of a moving target. It is a measure of how well the eye movement system keeps up with the speed of the moving object in the vertical plane. Specifically, gain is calculated as the ratio of eye movement velocity to target velocity. The participant sits in front of a computer screen displaying a moving symbol, which they must follow without moving their head. Eye movements are recorded and analyzed using an eye-tracking device.
Pupillometry - Amplitude | 1 year
  Pupillometry is the measurement and analysis of pupil size and its response to light stimuli. The amplitude i.e maximum constriction is the difference between the baseline pupil size and the smallest pupil size achieved after exposure to the light stimulus. The amplitude is measured in millimeters (mm).
Pupillometry - Velocity | 1 year
  Pupillometry is the measurement and analysis of pupil size and its response to light stimuli. The velocity is the speed at which the pupil constricts or dilates in response to changes in light intensity. Typically reported in millimeters per second (mm/s).

CONTACTS AND LOCATIONS:
Overall Officials: Nina Feddermann-Demont, PD Dr.med, Study Director — Medical Director

REFERENCES:
- [Background] Aderman MJ, Meister MR, Roach MH, Dengler BA, Ross JD, Malvasi SR, Cameron KL. Normative Values for Pupillary Light Reflex Metrics Among Healthy Service Academy Cadets. Mil Med. 2024 Jul 3;189(7-8):1593-1602. doi: 10.1093/milmed/usad271. PMID 37522744
- [Background] Brunner R, Bizzini M, Niedermann K, Maffiuletti NA. Epidemiology of Traumatic and Overuse Injuries in Swiss Professional Male Ice Hockey Players. Orthop J Sports Med. 2020 Oct 19;8(10):2325967120964720. doi: 10.1177/2325967120964720. eCollection 2020 Oct. PMID 33178879
- [Background] Chou TY, Huang YL, Leung W, Brown CN, Kaminski TW, Norcross MF. Does prior concussion lead to biomechanical alterations associated with lateral ankle sprain and anterior cruciate ligament injury? A systematic review and meta-analysis. Br J Sports Med. 2023 Dec;57(23):1509-1515. doi: 10.1136/bjsports-2023-106980. Epub 2023 Aug 30. PMID 37648411
- [Background] Clark JF, Ellis JK, Bench J, Khoury J, Graman P. High-performance vision training improves batting statistics for University of Cincinnati baseball players. PLoS One. 2012;7(1):e29109. doi: 10.1371/journal.pone.0029109. Epub 2012 Jan 19. PMID 22276103
- [Background] Clarsen B, Myklebust G, Bahr R. Development and validation of a new method for the registration of overuse injuries in sports injury epidemiology: the Oslo Sports Trauma Research Centre (OSTRC) overuse injury questionnaire. Br J Sports Med. 2013 May;47(8):495-502. doi: 10.1136/bjsports-2012-091524. Epub 2012 Oct 4. PMID 23038786
- [Background] Collins MW, Kontos AP, Reynolds E, Murawski CD, Fu FH. A comprehensive, targeted approach to the clinical care of athletes following sport-related concussion. Knee Surg Sports Traumatol Arthrosc. 2014 Feb;22(2):235-46. doi: 10.1007/s00167-013-2791-6. Epub 2013 Dec 12. PMID 24337463
- [Background] Covassin T, Elbin RJ. The female athlete: the role of gender in the assessment and management of sport-related concussion. Clin Sports Med. 2011 Jan;30(1):125-31, x. doi: 10.1016/j.csm.2010.08.001. PMID 21074087
- [Background] Covassin T, Savage JL, Bretzin AC, Fox ME. Sex differences in sport-related concussion long-term outcomes. Int J Psychophysiol. 2018 Oct;132(Pt A):9-13. doi: 10.1016/j.ijpsycho.2017.09.010. Epub 2017 Sep 18. PMID 28927725
- [Background] Dannenbaum E, Chilingaryan G, Fung J. Visual vertigo analogue scale: an assessment questionnaire for visual vertigo. J Vestib Res. 2011;21(3):153-9. doi: 10.3233/VES-2011-0412. PMID 21558640
- [Background] Domenech MA, Sizer PS, Dedrick GS, McGalliard MK, Brismee JM. The deep neck flexor endurance test: normative data scores in healthy adults. PM R. 2011 Feb;3(2):105-10. doi: 10.1016/j.pmrj.2010.10.023. PMID 21333948
- [Background] Eagle SR, Ferris LM, Mucha A, Sinnott A, Marchetti G, Trbovich A, Port N, Clugston J, Ortega J, Collins MW, Broglio SP, McAllister T, McCrea MA, Pasquina P, Kontos AP, Investigators CC. Minimum detectable change and false positive rates of the vestibular/ocular motor screening (VOMS) tool: an NCAA-DoD care consortium analysis. Brain Inj. 2021 Nov 10;35(12-13):1563-1568. doi: 10.1080/02699052.2021.1973561. Epub 2021 Sep 20. PMID 34543099
- [Background] Echemendia RJ, Brett BL, Broglio S, Davis GA, Giza CC, Guskiewicz KM, Harmon KG, Herring S, Howell DR, Master C, McCrea M, Naidu D, Patricios JS, Putukian M, Walton SR, Schneider KJ, Burma JS, Bruce JM. Sport concussion assessment tool - 6 (SCAT6). Br J Sports Med. 2023 Jun;57(11):622-631. doi: 10.1136/bjsports-2023-107036. No abstract available. PMID 37316203
- [Background] Eliason PH, Galarneau JM, Kolstad AT, Pankow MP, West SW, Bailey S, Miutz L, Black AM, Broglio SP, Davis GA, Hagel BE, Smirl JD, Stokes KA, Takagi M, Tucker R, Webborn N, Zemek R, Hayden A, Schneider KJ, Emery CA. Prevention strategies and modifiable risk factors for sport-related concussions and head impacts: a systematic review and meta-analysis. Br J Sports Med. 2023 Jun;57(12):749-761. doi: 10.1136/bjsports-2022-106656. PMID 37316182
- [Background] Emery CA, Cassidy JD, Klassen TP, Rosychuk RJ, Rowe BH. Effectiveness of a home-based balance-training program in reducing sports-related injuries among healthy adolescents: a cluster randomized controlled trial. CMAJ. 2005 Mar 15;172(6):749-54. doi: 10.1503/cmaj.1040805. PMID 15767608
- [Background] Faude O, Rossler R, Junge A, Aus der Funten K, Chomiak J, Verhagen E, Beaudouin F, Dvorak J, Feddermann-Demont N. Head injuries in children's football-results from two prospective cohort studies in four European countries. Scand J Med Sci Sports. 2017 Dec;27(12):1986-1992. doi: 10.1111/sms.12839. Epub 2017 Feb 3. PMID 28054391
- [Background] Feddermann-Demont N, Chiampas G, Cowie CM, Meyer T, Nordstrom A, Putukian M, Straumann D, Kramer E. Recommendations for initial examination, differential diagnosis, and management of concussion and other head injuries in high-level football. Scand J Med Sci Sports. 2020 Oct;30(10):1846-1858. doi: 10.1111/sms.13750. Epub 2020 Jun 29. PMID 32557913
- [Background] Feddermann-Demont N, Echemendia RJ, Schneider KJ, Solomon GS, Hayden KA, Turner M, Dvorak J, Straumann D, Tarnutzer AA. What domains of clinical function should be assessed after sport-related concussion? A systematic review. Br J Sports Med. 2017 Jun;51(11):903-918. doi: 10.1136/bjsports-2016-097403. PMID 29098983
- [Background] Feddermann-Demont N, Straumann D, Dvorak J. Return to play management after concussion in football: recommendations for team physicians. J Sports Sci. 2014;32(13):1217-28. doi: 10.1080/02640414.2014.918273. Epub 2014 Jun 6. PMID 24902964
- [Background] Gualtieri CT, Johnson LG. Reliability and validity of a computerized neurocognitive test battery, CNS Vital Signs. Arch Clin Neuropsychol. 2006 Oct;21(7):623-43. doi: 10.1016/j.acn.2006.05.007. Epub 2006 Oct 2. PMID 17014981
- [Background] Hanni S, Vedung F, Tegner Y, Marklund N, Johansson J. Soccer-Related Concussions Among Swedish Elite Soccer Players: A Descriptive Study of 1,030 Players. Front Neurol. 2020 Sep 23;11:510800. doi: 10.3389/fneur.2020.510800. eCollection 2020. PMID 33071939
- [Background] Jafarzadehpur E, Aazami N, Bolouri B. Comparison of saccadic eye movements and facility of ocular accommodation in female volleyball players and non-players. Scand J Med Sci Sports. 2007 Apr;17(2):186-90. doi: 10.1111/j.1600-0838.2005.00535.x. PMID 17394481
- [Background] Johnston W, O'Reilly M, Duignan C, Liston M, McLoughlin R, Coughlan GF, Caulfield B. Association of Dynamic Balance With Sports-Related Concussion: A Prospective Cohort Study. Am J Sports Med. 2019 Jan;47(1):197-205. doi: 10.1177/0363546518812820. Epub 2018 Dec 3. PMID 30501391
- [Background] Jorge J, Fernandes P. Static and dynamic visual acuity and refractive errors in elite football players. Clin Exp Optom. 2019 Jan;102(1):51-56. doi: 10.1111/cxo.12812. Epub 2018 Jul 28. PMID 30054950
- [Background] Kontos AP, Eagle SR, Chrisman SPD, Putukian M, Manderino L, Holland C, Collins MW, Broglio SP, McAllister TW, McCrea MA, Pasquina P, Kaminski TW; CARE Consortium Investigators. Incidence of concussion and associated risk factors in collegiate soccer: findings from the NCAA-DoD CARE consortium. Sci Med Footb. 2024 Aug;8(3):189-195. doi: 10.1080/24733938.2023.2227134. Epub 2023 Jun 23. PMID 37338928
- [Background] Kontos AP, Eagle SR, Mucha A, Kochick V, Reichard J, Moldolvan C, Holland CL, Blaney NA, Collins MW. A Randomized Controlled Trial of Precision Vestibular Rehabilitation in Adolescents following Concussion: Preliminary Findings. J Pediatr. 2021 Dec;239:193-199. doi: 10.1016/j.jpeds.2021.08.032. Epub 2021 Aug 25. PMID 34450120
- [Background] Lavigne A, Lamontagne M, Mares C, Gagnon DH. Ease of Use and Usefulness of a Newly Developed Mobile App to Monitor Pain and Adherence Among Individuals With an Achilles Tendinopathy Engaged in a Rehabilitation Program. Clin J Sport Med. 2023 Nov 1;33(6):e186-e189. doi: 10.1097/JSM.0000000000001184. Epub 2023 Aug 1. PMID 37526499
- [Background] Ling DI, Hannafin JA, Prather H, Skolnik H, Chiaia TA, de Mille P, Lewis CL, Casey E. The Women's Soccer Health Study: From Head to Toe. Sports Med. 2023 Oct;53(10):2001-2010. doi: 10.1007/s40279-023-01860-x. Epub 2023 May 17. PMID 37195359
- [Background] Makdissi M, Schneider KJ, Feddermann-Demont N, Guskiewicz KM, Hinds S, Leddy JJ, McCrea M, Turner M, Johnston KM. Approach to investigation and treatment of persistent symptoms following sport-related concussion: a systematic review. Br J Sports Med. 2017 Jun;51(12):958-968. doi: 10.1136/bjsports-2016-097470. Epub 2017 May 8. PMID 28483928
- [Background] Mandelbaum BR, Silvers HJ, Watanabe DS, Knarr JF, Thomas SD, Griffin LY, Kirkendall DT, Garrett W Jr. Effectiveness of a neuromuscular and proprioceptive training program in preventing anterior cruciate ligament injuries in female athletes: 2-year follow-up. Am J Sports Med. 2005 Jul;33(7):1003-10. doi: 10.1177/0363546504272261. Epub 2005 May 11. PMID 15888716
- [Background] McCrory P, Meeuwisse WH, Dvorak J, Echemendia RJ, Engebretsen L, Feddermann-Demont N, McCrea M, Makdissi M, Patricios J, Schneider KJ, Sills AK. 5th International Conference on Concussion in Sport (Berlin). Br J Sports Med. 2017 Jun;51(11):837. doi: 10.1136/bjsports-2017-097878. No abstract available. PMID 29098980
- [Background] Mihalik JP, Teel EF, Ford CB, Amalfe SA, Barczak-Scarboro NE, Lynall RC, Riegler KE, Wasserman EB, Putukian M. The Effect of Sex, Sport, and Preexisting Histories on Baseline Concussion Test Performance in College Lacrosse and Soccer Athletes. Clin J Sport Med. 2022 Sep 1;32(5):e461-e468. doi: 10.1097/JSM.0000000000001018. Epub 2022 Feb 15. PMID 36083332
- [Background] Morelli N, Heebner NR, DeFeo CJ, Hoch MC. The Influence of Cognitive Dual Tasks on Concussion Balance Test Performance. Motor Control. 2021 Feb 8;25(2):252-263. doi: 10.1123/mc.2020-0075. PMID 33567406
- [Background] Mucci V, Meier C, Bizzini M, Romano F, Agostino D, Ventura A, Bertolini G, Feddermann-Demont N. Combined Optokinetic Treatment and Vestibular Rehabilitation to Reduce Visually Induced Dizziness in a Professional Ice Hockey Player After Concussion: A Clinical Case. Front Neurol. 2019 Nov 29;10:1200. doi: 10.3389/fneur.2019.01200. eCollection 2019. PMID 31849804
- [Background] Orchard JW, Meeuwisse W, Derman W, Hagglund M, Soligard T, Schwellnus M, Bahr R. Sport Medicine Diagnostic Coding System (SMDCS) and the Orchard Sports Injury and Illness Classification System (OSIICS): revised 2020 consensus versions. Br J Sports Med. 2020 Apr;54(7):397-401. doi: 10.1136/bjsports-2019-101921. Epub 2020 Feb 29. PMID 32114487
- [Background] Ozinga SJ, Linder SM, Koop MM, Dey T, Figler R, Russman AN, So R, Rosenthal AH, Cruickshank J, Alberts JL. Normative Performance on the Balance Error Scoring System by Youth, High School, and Collegiate Athletes. J Athl Train. 2018 Jul;53(7):636-645. doi: 10.4085/1062-6050-129-17. Epub 2018 Aug 15. PMID 30109948
- [Background] Patricios JS, Schneider KJ, Dvorak J, Ahmed OH, Blauwet C, Cantu RC, Davis GA, Echemendia RJ, Makdissi M, McNamee M, Broglio S, Emery CA, Feddermann-Demont N, Fuller GW, Giza CC, Guskiewicz KM, Hainline B, Iverson GL, Kutcher JS, Leddy JJ, Maddocks D, Manley G, McCrea M, Purcell LK, Putukian M, Sato H, Tuominen MP, Turner M, Yeates KO, Herring SA, Meeuwisse W. Consensus statement on concussion in sport: the 6th International Conference on Concussion in Sport-Amsterdam, October 2022. Br J Sports Med. 2023 Jun;57(11):695-711. doi: 10.1136/bjsports-2023-106898. PMID 37316210
- [Background] Piras A, Lobietti R, Squatrito S. A study of saccadic eye movement dynamics in volleyball: comparison between athletes and non-athletes. J Sports Med Phys Fitness. 2010 Mar;50(1):99-108. PMID 20308980
- [Background] Prien A, Grafe A, Rossler R, Junge A, Verhagen E. Epidemiology of Head Injuries Focusing on Concussions in Team Contact Sports: A Systematic Review. Sports Med. 2018 Apr;48(4):953-969. doi: 10.1007/s40279-017-0854-4. PMID 29349651
- [Background] Quevedo-Junyent L, Aznar-Casanova JA, Merindano-Encina D, Cardona G, Sole-Forto J. Comparison of dynamic visual acuity between water polo players and sedentary students. Res Q Exerc Sport. 2011 Dec;82(4):644-51. doi: 10.1080/02701367.2011.10599801. PMID 22276406
- [Background] Soligard T, Myklebust G, Steffen K, Holme I, Silvers H, Bizzini M, Junge A, Dvorak J, Bahr R, Andersen TE. Comprehensive warm-up programme to prevent injuries in young female footballers: cluster randomised controlled trial. BMJ. 2008 Dec 9;337:a2469. doi: 10.1136/bmj.a2469. PMID 19066253
- [Background] Tarnutzer AA, Weber KP, Bockisch CJ, Straumann D, Feddermann-Demont N. Vestibular performance in high-level soccer and ice hockey players: Sport-specific norm values and implications. J Sci Med Sport. 2022 Jan;25(1):81-88. doi: 10.1016/j.jsams.2021.08.003. Epub 2021 Aug 13. PMID 34509343
- [Background] Truong JQ, Ciuffreda KJ. Comparison of pupillary dynamics to light in the mild traumatic brain injury (mTBI) and normal populations. Brain Inj. 2016;30(11):1378-1389. doi: 10.1080/02699052.2016.1195922. Epub 2016 Aug 19. PMID 27541745
- [Background] Truong JQ, Ciuffreda KJ. Quantifying pupillary asymmetry through objective binocular pupillometry in the normal and mild traumatic brain injury (mTBI) populations. Brain Inj. 2016;30(11):1372-1377. doi: 10.1080/02699052.2016.1192220. Epub 2016 Aug 11. PMID 27712127
- [Background] Vedung F, Hanni S, Tegner Y, Johansson J, Marklund N. Concussion incidence and recovery in Swedish elite soccer - Prolonged recovery in female players. Scand J Med Sci Sports. 2020 May;30(5):947-957. doi: 10.1111/sms.13644. Epub 2020 Mar 12. PMID 32100894
- [Background] Visscher RMS, Feddermann-Demont N, Romano F, Straumann D, Bertolini G. Artificial intelligence for understanding concussion: Retrospective cluster analysis on the balance and vestibular diagnostic data of concussion patients. PLoS One. 2019 Apr 2;14(4):e0214525. doi: 10.1371/journal.pone.0214525. eCollection 2019. PMID 30939164
- [Background] Walden M, Mountjoy M, McCall A, Serner A, Massey A, Tol JL, Bahr R, D'Hooghe M, Bittencourt N, Della Villa F, Dohi M, Dupont G, Fulcher M, Janse van Rensburg DCC, Lu D, Andersen TE. Football-specific extension of the IOC consensus statement: methods for recording and reporting of epidemiological data on injury and illness in sport 2020. Br J Sports Med. 2023 Nov;57(21):1341-1350. doi: 10.1136/bjsports-2022-106405. Epub 2023 Jan 6. PMID 36609352
- [Background] Weber ML, Lynall RC, Hoffman NL, Miller EH, Kaminski TW, Buckley TA, Benjamin HJ, Miles CM, Whitlow CT, Lintner L, Broglio SP, McCrea M, McAllister T, Schmidt JD; CARE Consortium Investigators. Health-Related Quality of Life Following Concussion in Collegiate Student-Athletes With and Without Concussion History. Ann Biomed Eng. 2019 Oct;47(10):2136-2146. doi: 10.1007/s10439-018-02151-7. Epub 2018 Oct 9. PMID 30302664
- [Background] Williams AM, Ward P, Chapman C. Training perceptual skill in field hockey: is there transfer from the laboratory to the field? Res Q Exerc Sport. 2003 Mar;74(1):98-103. doi: 10.1080/02701367.2003.10609068. No abstract available. PMID 12659480
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Attwood MJ, Roberts SP, Trewartha G, England ME, Stokes KA. Efficacy of a movement control injury prevention programme in adult men's community rugby union: a cluster randomised controlled trial. Br J Sports Med. 2018 Mar;52(6):368-374. doi: 10.1136/bjsports-2017-098005. Epub 2017 Oct 21. PMID 29055883